CLINICAL TRIAL: NCT01488110
Title: Undersökning av ny Behandlingsmetod Vid migränanfall (Evaluation of a New Treatment for Migraine Attacks)
Brief Title: Investigation of Efficacy and Outcome of a New Medical Device for Treatment of Migraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too slow recruitment rate. The study has been terminated and will be re-started with an improved and more suitable study design.
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jan-Erik Juto, Adjunct professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Migraine2011/1609-31/2
Record Dates: First submitted 2011-12-02; First posted 2011-12-08 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Migraine medical device (Experimental): Treatment with an active nasal probe
  Interventions: Device: In-house prototype invented by Jan-Erik Juto
- Inactive migraine medical device (Placebo Comparator): Treatment with an inactive nasal probe.
  Interventions: Device: In-house prototype invented by Jan-Erik Juto

INTERVENTIONS:
Device: In-house prototype invented by Jan-Erik Juto — 30 minutes treatment with an active nasal probe.
  Arms: Migraine medical device
Device: In-house prototype invented by Jan-Erik Juto — 30 minutes treatment with an inactive nasal probe.
  Arms: Inactive migraine medical device

SUMMARY:
The purpose of this study is to evaluate the efficacy of a novel therapy for treatment of migraine, pain reduction and relief of associated symptoms during ongoing migraine attacks, and presence of a preventive effect two months post treatment. Another purpose is to investigate if and how this treatment affects manifestations of the autonomic nervous system activity.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects, in otherwise good health, 20 to 55 years of age
* Subjects who meet the ICHD-2 (2nd Edition of The International Headache Classification) criteria for migraine headache
* Subjects with a minimum of 1 migraine attack per month
* Attack duration of 4 to 72 hours
* Normal attack intensity of at least 4 on a 0-10 VAS-scale

Exclusion Criteria:

* Completed heart surgery
* Cardiovascular diseases
* Vascular damages on neck vessels
* Diseases other than migraine of the CNS
* Severe disease of vital body organs
* Severe psychiatric disorders
* More than 6 migraine attacks per month

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01

PRIMARY OUTCOMES:
Change from baseline in pain intensity according to VAS-scales (0-10) | Estimation 40 minutes
  Documentation of pain intensity prior to treatment initiation (baseline value), every 5 minutes during treatment and post treatment.

SECONDARY OUTCOMES:
RR (Heart rate)-interval | Estimation 40 minutes
  ECG will be obtained during treatment
Change from baseline in sympathetic nervous system activity | Estimation 40 minutes
  Plethysmographic measurements will be obtained during treatment (finger clamp on finger).
Blood pressure | Estimation 40 minutes
  Will be obtained prior to treatment initiation and post treatment
Change from baseline in attack frequency based on completed patient diaries | 3 to 4 months
Change from baseline in attack intensity based on completed patient diaries | 3 to 4 months
Change from baseline in attack duration based on completed patient diaries | 3 to 4 months
Change from baseline in medicine consumption based on completed patient diaries | 3 to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Juto, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm, Sweden